CLINICAL TRIAL: NCT04673526
Title: Laparoscopic Intersphincteric Resection for Ultra Low Rectal Cancer in Elderly Patients: Oncological and Functional Lon Term Outcome. A Prospective Case Control Study.
Brief Title: Laparoscopic Intersphincteric Resection in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASL Verbano Cusio Ossola (Other Government)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marco Giacometti, Principal Investigator, ASL Verbano Cusio Ossola
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lap IRR 70+
Record Dates: First submitted 2020-11-19; First posted 2020-12-17 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Rectal Cancer
Keywords: intersphincteric resection; elderly; rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective case-control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intersphincteric resection (Experimental): After a laparoscopic TME (total mesorectal excision) is carried out down to the elevator ani plane and the anorectal junction, the intersphincteric plane is dissected, opening the space between puborectalis muscle and interior sphincter. Margin of resection is at least 1 cm below the lower margin of the tumor. Rectal excision is completed with transanal circumferential dissection and after specimen extraction through the anus, a colo-anal hand sewn anastomosis is fashioned.
  Interventions: Procedure: Laparoscopic intersphincteric resection
- Abdomen-perineal procedures (Active Comparator): After identification of the elevator ani plane, the descendent colon is transected with a linear stapler and a terminal stoma is fashioned. Then, a circumferential incision is made around anal orifice and perineal dissection is performed circumferentially to the pelvic cavity. Perineal defect is repaired performing mono-lateral or bilateral inferior gluteal flap.
  Interventions: Procedure: Laparoscopic abdomino-perineal procedures

INTERVENTIONS:
Procedure: Laparoscopic intersphincteric resection — Laparoscopic intersphincteric resection for ultra low rectal cancer in elderly patients
  Arms: Intersphincteric resection
Procedure: Laparoscopic abdomino-perineal procedures — Abdominoperineal resection + colostomy in left iliac fossa or perineum
  Arms: Abdomen-perineal procedures

SUMMARY:
The aim of the present study is to assess if it is possible to offer intersphincteric rectal resection (IRR) to selected patients older than 70 years affected by ultra-low rectal cancer. The study, involving patients with rectal cancer at less than 5 cm from the anal verge, will compare elderly patients refusing standard sphincteric demolition and undergoing IRR, with some control groups (younger patients undergoing IRR, >70 years old patients undergoing abdominoperineal resection + colostomy in left iliac fossa, >70 years old patients undergoing abdominoperineal resection + perineal colostomy). The groups will be compared in terms of quality of life, quality of life associated to incontinence, overall survival, disease free survival and post-operative complications. This will be helpful to identify conditions for extending IRR to elderly patients. The study is run by Colo-rectal Surgery Unit at Policlinico San Matteo in Pavia (Italy) from 2009 to 2016, directly led by Dr. Sandro Zonta (principal investigator) and funded by the hospital itself.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years old who were affected by rectal cancer sited lower than 5 cm from anal verge and refused abdomen-perineal treatment.

Exclusion Criteria:

* Cancer extension over internal sphincteric muscle (T4) evaluated through MRI during staging work out;
* diabetic neuropathy conditioning previous partial/total incontinence;
* other pre-existing pathological condition affecting faecal incontinence.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of life of operated patients as assessed by Quality of Life Short Form Health Survey (QoL SF-36) | 6 months after discharge
  QoL SF-36 score (Quality of Life Short Form Health Survey from 0 to 100, with the lower score the more disability)
Quality of life associated to incontinence as assessed by Wexner incontinence score (WiS) | 6 months after discharge
  WiS (Wexner incontinence score) from 0 to 20: higher score means worse incontinence
Quality of life associated to incontinence as assessed by Faecal incontinence quality of life scale (FIQL) | 6 months after discharge
  FIQL (Faecal incontinence quality of life scale): 29 items from 1 to 6 - the lower value the worse quality of life

SECONDARY OUTCOMES:
Patients' survival | 5 years
  months
Disease free survival | 5 years
  months
Post-operative complications | 6 months after discharge
  Clavien-Dindo score from grade I (minor complications) to grade V (death)

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Zonta, PhD, Principal Investigator — ASL VCO
Locations (1):
- Sandro Zonta, Domodossola, VCO, Italy

IPD SHARING:
Plan to Share IPD: No